CLINICAL TRIAL: NCT02854956
Title: Clinical Phenotyping and Characterization of Neural Networks and Cognitive Processes Involved in Mental Retardation X-linked
Acronym: XLMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2010-609
Record Dates: First submitted 2016-06-29; First posted 2016-08-04 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: X-linked Mental Retardation
Keywords: phenotype; X-linked mental retardation; neuronal networks; cognitive processes
MeSH Terms: conditions — X-Linked Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- X-linked Mental retardation (Other): This is an observational study which will allow to precisely describe the phenotype associated to each X-linked mental retardation gene.
  Interventions: Behavioral: Neuropsychological, cognitive and behavioral assessment
- Control Group (Other): This group will be compared to X-linked mental retardation group in order to obtain a baseline on some cognitive tests.
  Interventions: Behavioral: Neuropsychological, cognitive and behavioral assessment

INTERVENTIONS:
Behavioral: Neuropsychological, cognitive and behavioral assessment — The assessment includes mainly :
  * The Raven's Progressives matrices test which allow to assess the non-verbal reasoning mental age of the patient
  * The Wechsler scale or Brunet Lézine scale which allow to assess The Intellectual Quotient
  * The Peabody Picture Vocabulary Test Revised which allow to determine the Vocabulary age (receptive language).
  * The Vineland adaptive behavioral scale which allow to assess the adaptive behavior
  * The Nisonger child behavior rating form which allow to assess the behavior disorders
  * Analogical visual reasoning task (eye-tracking assessment and behavior assessment) which allow to identify the strategy used to solve the task and provides an objective and quantitative assessment of visual analogical reasoning and cognitive inhibition.
  * Kinematic analysis of a grasping movement which allow to study the effect of the orientation and the type of pinch on the movement duration and both the transport component and the grasp component.

SUMMARY:
X-linked Mental retardation (XLMR) represent 10% of the causes of mental retardation with a prevalence in both sexes around 1/296, i.e. 3.3 / 1000 births (Opitz et al., 1986). This heterogeneous group of XLMR includes dozens of rare diseases, some of them affecting only a few patients. Molecular diagnosis is currently available in France for 25 XLMR genes, within the national network of XLMR molecular diagnosis. However, whereas some syndromes such as Fragile X syndrome, are now well clinically defined, this is not the case for recently identified syndromes for which very few data is available, preventing clinicians to focus molecular diagnosis on a specific gene.

Therefore, this study aims to :

* Achieve a description of the clinical phenotype specific to each XLMR gene (Phase 1 of the study, n=200)
* Characterize the cognitive learning mechanisms and dysfunctional neural networks involved (Phase 2 of the study, n=75, i.e. 5 groups of 15 patients with a mutation in the same gene). These two elements constitute key steps to develop appropriate rehabilitation strategies and targeted pharmacological therapies.

Moreover, the impact of mental retardation on the primary caregiver within the family and the induced burden in terms of psycho-social, organizational and economic burden will also be assessed. These elements, directly related to the patient's environment, are very important to characterize in order to better understand the consequences of each gene mutation (Phase 3 of the study, n=283). For example, it is necessary to better understand the impact of Fragile X syndrome in terms of capacity and behavior, lifestyle, and health care needs of the patients While advancing knowledge allows to consider innovative therapeutics, the implementation of these therapeutics and assessment of their impact on the patients' life trajectory, require precise characterization of the population to be treated in medico socioeconomic terms.

ELIGIBILITY:
Inclusion Criteria:

* Age : from 2 to 60 years old
* Having a pathogenic mutation of one of the X chromosome genes associated with :

  * For boys : mental retardation (IQ<70), and/or developmental delay (DQ<70) and/or pervasive developmental disorder (autism, Asperger…)
  * For girls : mental retardation (IQ<70), and/or developmental delay (DQ<70) and/or pervasive developmental disorder (autism, Asperger…) and/or specific learning disabilities

Exclusion Criteria:

* patient or parents refusal to participate in the study
* genetic polymorphism in a X chromosome gene involved in mental retardation but not considered as pathogenic
* person refusing to be informed if an abnormality would be discovered during medical examination

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 573 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-12 (Actual); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotyping of neurodevelopment: acquisition age of early developmental skills (motor and language), and the adaptive skills profile (Vineland adaptive behavioral scale) | at inclusion (Day 1)
  The primary outcome measure is composite and includes acquisition age of early developmental skills (motor and language), and the adaptive skills profile (Vineland adaptive behavioral scale). The Vineland adaptive behavioral scale performed during a semi-structured interview of the parents of the patient, will assess the adaptive behavior profile of the patient (including communication, daily living skills, socialization, motricity and the global adaptive score).

SECONDARY OUTCOMES:
Intellectual functioning assessment (Wechsler scale) | at inclusion (Day 1)
  The Intellectual Quotient of the patient will be assessed using a Wechsler scale, adapted to the age of the patient. For patients younger than 3 years or too severely impaired to perform a Wechsler scale, the Brunet Lézine scale will be used.
Raven's Progressive matrices | at inclusion (Day 1)
  The Raven's Progressives matrices test will allow to assess the non-verbal reasoning mental age of the patient
Peabody Picture Vocabulary Test Revised | at inclusion (Day 1)
  The Peabody Picture Vocabulary Test Revised will allow to determine the Vocabulary age (receptive language) of the patient.
Edinburgh handedness test | at inclusion (Day 1)
  The Edinburgh handedness test will assess the handedness of the patients.
Birth parameters: weight, height and head circumference and APGAR score | at inclusion (Day 1)
  The birth parameters include weight, height and head circumference at birth, as well as the initial cardiac and pulmonary adaptation (APGAR score).
Nisonger child behavior rating form | at inclusion (Day 1)
  The Nisonger child behavior rating form will allow the assessment of behavior disorders including: conduct disorders, anxiety, hyperactivity, automutilation/stereotyped behavior, self-isolation/rituals, sensitivity/susceptibility.
Caregiver Burden Inventory Modified | at inclusion (Day 1)
  The Caregiver Burden Inventory Modified will allow the assessment of the impact of mental retardation on the primary caregiver within the family.
Analogical visual reasoning task (behavior assessment) | at inclusion (Day 1)
  This paradigm (HCL/CNRS patented), appropriate for mentally retarded patients provides an objective and quantitative assessment of visual analogical reasoning and cognitive inhibition.
Analogical visual reasoning task (eye-tracking assessment) | at inclusion (Day 1)
  The eye-tracking analysis of this paradigm (HCL/CNRS patented) made it possible to identify the strategy used by participants to solve the task. Mentally Retarded patients are not able to explicitly explain the strategy they used to solve the task, but with eye-tracking analysis, we can understand how they performed the task, which is crucial information in order to help them improve their performance through remediation strategies.
Kinematic analysis of a grasping movement | at inclusion (Day 1)
  This kinematic analysis of a grasping movement will allow us to study the effect of the orientation (+56°or -56°) and the type of pinch (thumb-index, thumb-middle finger and thumb-annular) on the movement duration and both the transport component (wrist acceleration and velocity peaks, latencies and amplitudes) and the grasp component (maximum grip aperture latency and amplitude and opposition axis).
Structural neuroimaging by MRI | at inclusion (Day 1)
  Structural brain MRI analysis will determine if a specific morphological neuroanatomical pattern can be found for each X-linked mental retardation gene.
Functional neuroimaging by MRI | at inclusion (Day 1)
  Functional brain MRI analysis will determine if patients with X-linked mental retardation have a specific functional neuroanatomical pattern associated to the reasoning task.
School curriculum: age and type of shool | at inclusion (Day 1)
  The school curriculum will include the age at school entrance, and the type of school the child went to.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DESPORTES, Pr, Principal Investigator — Groupement Hospitalier Est - Hôpital Femme Mère Enfant - Service de neurologie pédiatrique
Locations (1):
- Groupement Hospitalier Est - Hôpital Femme Mère Enfant - Service de neurologie pédiatrique, Bron, France